CLINICAL TRIAL: NCT06611033
Title: A Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of V118 Formulation C in Healthy Adults
Brief Title: A Study of V118 Formulation C (V118C) in Healthy Participants (V118C-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: V118C-001
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- V118C (Experimental): Participants receive intramuscular (IM) injection of V118C in a 2-dose regimen administered on Day 1 and Day 29.
  Interventions: Biological: V118C
- V118 (Experimental): Participants receive IM injection of V118 in a 2-dose regimen administered on Day 1 and Day 29.
  Interventions: Biological: V118; Biological: Saline
- PREVNAR 20™ + Saline (Active Comparator): Participants receive one dose of IM injection of PREVNAR 20™ in a 2-dose regimen on Day 1 followed by one dose of saline on Day 29.
  Interventions: Biological: PREVNAR 20™; Biological: Saline

INTERVENTIONS:
Biological: V118C — Intramuscular Administration
  Arms: V118C
Biological: V118 — Intramuscular Administration
  Arms: V118
Biological: PREVNAR 20™ — Intramuscular Administration
  Arms: PREVNAR 20™ + Saline
Biological: Saline — Intramuscular Administration
  Arms: PREVNAR 20™ + Saline; V118

SUMMARY:
The goal of this study is to learn how safe V118 Formulation C is in Healthy Adults and how well people tolerate it.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Is in good health before randomization

Exclusion Criteria:

* Has a history of invasive pneumococcal disease or known history of other culture-positive pneumococcal disease within 3 years prior to receiving study vaccination.
* Has a history of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Injection Site Adverse Events (AEs) | Up to approximately 7 days after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants with a solicited injection-site AE will be reported.
Number of Participants with Solicited Systemic AEs | Up to approximately 7 days after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants with a solicited systemic AE will be reported.
Number of Participants with Immediate AEs Following Vaccination | Up to approximately 30 minutes after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants with Immediate AEs following vaccination will be reported.
Number of Participants with Unsolicited AEs | Up to approximately 28 days after each vaccination
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. An unsolicited AE is an AE that is not solicited using a vaccine report card (VRC) and that is communicated by a participant. The number of participants that experienced an unsolicited AE will be reported.
Number of Participants With a Serious Adverse Event (SAE) | Up to approximately 12 months after final vaccination
  An SAE is defined as any untoward medical occurrence that at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. The number of participants who experience an SAE will be reported.
Number of Participants with a Medically Attended Adverse Event (MAAE) | Up to approximately 12 months after final vaccination
  An MAAE is defined as an adverse event in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency room visit, office visit, or an urgent care visit with any medical personnel for any reason. The number of participants who experience an MAAE will be reported.
Number of Participants with an Event of Clinical Interest (ECI) | Up to approximately 12 months after final vaccination
  An ECI includes but is not limited to: 1) An overdose defined as: A participant receiving more than 1 dose of study vaccine in a 24-hour period or more than 2 doses of study vaccine throughout the study. 2) Potential drug-induced liver injury (DILI) events defined as: An elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) lab value that is ≥3 times the upper limit of normal (ULN) and an elevated total bilirubin lab value that is ≥2 times ULN and, at the same time, an alkaline phosphatase lab value that is <2 times ULN, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing. 3) Potential immune-mediated disease (pIMDs) defined as: A subset of AEs that include either an established autoimmune disease(s) or Inflammatory and/or neurologic disorder(s), which might or might not have an autoimmune etiology. The number of participants who experience an ECI will be reported.

SECONDARY OUTCOMES:
Serotype-specific Immunoglobulin G (IgG) geometric mean concentrations (GMCs) | Day 28 postvaccination
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Velocity Clinical Research, Hallandale Beach ( Site 0003), Hallandale, Florida
  - Research Centers of America ( Hollywood ) ( Site 0002), Hollywood, Florida
  - University of Texas Medical Branch ( Site 0001), Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com